CLINICAL TRIAL: NCT00118404
Title: Prophylactic Cognitive Therapy for Depression.
Brief Title: Cognitive Therapy for Recurrent Depression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Robin Jarrett, Professor of Psychiatry, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R01MH058397 (NIH); R01MH058397 (NIH); R01MH069619 (NIH); R01MH058356 (NIH); R01MH069618 (NIH); NCT00183664 (obsolete NCT alias); NCT00218764 (obsolete NCT alias)
Record Dates: First submitted 2005-07-06; First posted 2005-07-11 (Estimated); Results first posted 2014-06-05 (Estimated); Last update posted 2014-06-05 (Estimated); Status verified 2014-05

CONDITIONS: Depression
Keywords: Cognitive therapy; Antidepressants; Psychotherapy
MeSH Terms: conditions — Depression | interventions — Fluoxetine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Participants received acute phase and continuation phase cognitive therapy
  Interventions: Behavioral: Continuation phase cognitive therapy; Behavioral: Acute phase cognitive therapy
- 2 (Placebo Comparator): Participants received acute phase cognitive therapy and continuation phase pill placebo
  Interventions: Other: Continuation phase pill placebo; Behavioral: Acute phase cognitive therapy
- 3 (Active Comparator): Participants received acute phase cognitive therapy and continuation phase fluoxetine
  Interventions: Drug: Continuation phase fluoxetine; Behavioral: Acute phase cognitive therapy

INTERVENTIONS:
Behavioral: Continuation phase cognitive therapy — Continuation phase cognitive therapy included 10 sessions over 8 months.
  Arms: 1
Drug: Continuation phase fluoxetine — The dosage of fluoxetine was increased to 40 mg over 8 months.
  Other Names: Prozac
  Arms: 3
Other: Continuation phase pill placebo — The dosage of pill placebo was increased to 40 mg over 8 months.
  Arms: 2
Behavioral: Acute phase cognitive therapy — For the first 12 weeks, all participants received between 16 and 20 cognitive therapy sessions.

SUMMARY:
This study determined the effectiveness of continuation phase cognitive therapy versus antidepressant medication in preventing relapse of depression in people with recurrent depression.

DETAILED DESCRIPTION:
Cognitive therapy (CT) is a short-term talking therapy that focuses on changing negative thinking patterns and helping patients develop coping skills to deal with their experiences. Evidence suggests that CT is effective in treating a number of psychiatric conditions, including anxiety and anger. This study will determine the effectiveness of cognitive therapy versus antidepressant medication or placebo in preventing relapse of depression in people with recurrent depression.

This study lasted approximately 36 months and comprised three phases. For the first 12 weeks, all participants received between 16 and 20 CT sessions. Participants were then randomly assigned to receive additional CT sessions, antidepressants, or placebo for an additional 8 months. Upon completing treatment, participants entered follow-up study visits once every 4 months for the next 24 months. Clinician-rated scales and questionnaires were used to assess depressive symptoms of participants at study start and at the end of each study phase.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent unipolar major depressive disorder
* Have experienced at least two episodes of major depression
* Have experienced at least one period of recovery during a depressive episode or have a history of dysthymia (a mood disorder characterized by depression) prior to the onset of current or past depressive episodes
* Willing and able to comply with all study requirements
* Able to speak and read English

Exclusion Criteria:

* Active alcohol or other substance dependence within 6 months prior to study entry
* Currently at risk for suicide
* Mood disorders due to a medical condition or substance abuse
* Bipolar, schizoaffective, obsessive compulsive, or eating disorders
* Schizophrenia
* Unable to stop mood-altering medications
* Current use of medication or diagnosis of a medical disorder that may cause depression (e.g., diabetes, head injury, stroke, cancer, multiple sclerosis)
* Previous failure to experience a reduction in depressive symptoms after 8 weeks of cognitive therapy with a certified therapist
* Previous failure to experience a reduction in depressive symptoms after 6 weeks of 40 mg of Prozac
* Pregnancy or plan to become pregnant in the next 11-12 months
* Unable to attend clinic twice weekly during business hours
* Unable to complete questionnaires

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 523 (Actual)
Dates: Start 2000-03; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robin B. Jarrett, PhD, Principal Investigator — University of Texas, Southwestern Medical Center at Dallas
Locations (2):
- United States (2):
  - University of Pittsburgh Medical Center Western Psychiatric Institute and Clinic, Pittsburgh, Pennsylvania
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas

REFERENCES:
- [Background] Jarrett RB, Thase ME. Comparative efficacy and durability of continuation phase cognitive therapy for preventing recurrent depression: design of a double-blinded, fluoxetine- and pill placebo-controlled, randomized trial with 2-year follow-up. Contemp Clin Trials. 2010 Jul;31(4):355-77. doi: 10.1016/j.cct.2010.04.004. Epub 2010 May 6. PMID 20451668
- [Result] Jarrett RB, Vittengl JR, Clark LA, Thase ME. Skills of Cognitive Therapy (SoCT): a new measure of patients' comprehension and use. Psychol Assess. 2011 Sep;23(3):578-86. doi: 10.1037/a0022485. PMID 21319902
- [Result] Dunn TW, Vittengl JR, Clark LA, Carmody T, Thase ME, Jarrett RB. Change in psychosocial functioning and depressive symptoms during acute-phase cognitive therapy for depression. Psychol Med. 2012 Feb;42(2):317-26. doi: 10.1017/S0033291711001279. Epub 2011 Jul 25. PMID 21781377
- [Result] Smits JA, Minhajuddin A, Thase ME, Jarrett RB. Outcomes of acute phase cognitive therapy in outpatients with anxious versus nonanxious depression. Psychother Psychosom. 2012;81(3):153-60. doi: 10.1159/000334909. Epub 2012 Mar 3. PMID 22398963
- [Result] Renner F, Jarrett RB, Vittengl JR, Barrett MS, Clark LA, Thase ME. Interpersonal problems as predictors of therapeutic alliance and symptom improvement in cognitive therapy for depression. J Affect Disord. 2012 May;138(3):458-67. doi: 10.1016/j.jad.2011.12.044. Epub 2012 Feb 4. PMID 22306232
- [Result] Jarrett RB, Minhajuddin A, Borman PD, Dunlap L, Segal ZV, Kidner CL, Friedman ES, Thase ME. Cognitive reactivity, dysfunctional attitudes, and depressive relapse and recurrence in cognitive therapy responders. Behav Res Ther. 2012 May;50(5):280-6. doi: 10.1016/j.brat.2012.01.008. Epub 2012 Feb 21. PMID 22445946
- [Result] Brandon AR, Minhajuddin A, Thase ME, Jarrett RB. Impact of reproductive status and age on response of depressed women to cognitive therapy. J Womens Health (Larchmt). 2013 Jan;22(1):58-66. doi: 10.1089/jwh.2011.3427. PMID 23305218
- [Result] Jarrett RB, Minhajuddin A, Kangas JL, Friedman ES, Callan JA, Thase ME. Acute phase cognitive therapy for recurrent major depressive disorder: who drops out and how much do patient skills influence response? Behav Res Ther. 2013 May;51(4-5):221-30. doi: 10.1016/j.brat.2013.01.006. PMID 23485420
- [Result] Jarrett RB, Minhajuddin A, Gershenfeld H, Friedman ES, Thase ME. Preventing depressive relapse and recurrence in higher-risk cognitive therapy responders: a randomized trial of continuation phase cognitive therapy, fluoxetine, or matched pill placebo. JAMA Psychiatry. 2013 Nov;70(11):1152-60. doi: 10.1001/jamapsychiatry.2013.1969. PMID 24005123
- [Result] Vittengl JR, Clark LA, Thase ME, Jarrett RB. Nomothetic and idiographic symptom change trajectories in acute-phase cognitive therapy for recurrent depression. J Consult Clin Psychol. 2013 Aug;81(4):615-26. doi: 10.1037/a0032879. Epub 2013 Apr 29. PMID 23627652
- [Result] Vittengl JR, Clark LA, Thase ME, Jarrett RB. Replication and extension: separate personality traits from states to predict depression. J Pers Disord. 2014 Apr;28(2):225-46. doi: 10.1521/pedi_2013_27_117. Epub 2013 Jun 20. PMID 23786268
- [Derived] Callan JA, Kazantzis N, Park SY, Moore CG, Thase ME, Minhajuddin A, Kornblith S, Siegle GJ. A Propensity Score Analysis of Homework Adherence-Outcome Relations in Cognitive Behavioral Therapy for Depression. Behav Ther. 2019 Mar;50(2):285-299. doi: 10.1016/j.beth.2018.05.010. Epub 2018 Jun 5. PMID 30824246
- [Derived] Brown GK, Thase ME, Vittengl JR, Borman PD, Clark LA, Jarrett RB. Assessing cognitive therapy skills comprehension, acquisition, and use by means of an independent observer version of the Skills of Cognitive Therapy (SoCT-IO). Psychol Assess. 2016 Feb;28(2):205-13. doi: 10.1037/pas0000080. Epub 2015 Sep 7. PMID 26348032
- [Derived] Horner MS, Siegle GJ, Schwartz RM, Price RB, Haggerty AE, Collier A, Friedman ES. C'mon get happy: reduced magnitude and duration of response during a positive-affect induction in depression. Depress Anxiety. 2014 Nov;31(11):952-60. doi: 10.1002/da.22244. Epub 2014 Mar 18. PMID 24643964
- See also: Psychosocial Research and Depression Clinic — http://www.utsouthwestern.edu/utsw/home/research/prdc/indec.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult outpatients diagnosed with recurrent major depressive disorder (MDD) using the Structured Clinical Interview for Diagnostic and Statistical Manual-IV were recruited from January 2000-July 2008. The first diagnostic evaluation was completed in March 2000.
Pre-assignment Details: Eligible patients (n=523) entered 12-14 weeks of acute phase cognitive therapy. Responders (no MDD & Hamilton Rating Scale for Depression [HRSD] ≤12) were divided by lower & higher risk based on the final 7 HRSD scores. Only consenting, higher risk patients (N=241) were randomized into the 3 arms below. See Jarrett &Thase (2010) for design details.
Groups:
- Continuation Phase Fluoxetine: Participants received acute phase cognitive therapy and continuation phase pill placebo
  Acute phase cognitive therapy : For the first 12 weeks, all participants received between 16 and 20 cognitive therapy sessions.
  Continuation phase pill placebo : The dosage of pill placebo was increased to 40 mg over 8 months.
- Continuation Phase Cognitive Therapy: Participants received acute phase and continuation phase cognitive therapy
  Acute phase cognitive therapy : For the first 12 weeks, all participants received between 16 and 20 cognitive therapy sessions.
  Continuation phase cognitive therapy : Continuation phase cognitive therapy included 10 sessions over 8 months.
- Continuation Phase Pill Placebo: Participants received acute phase cognitive therapy and continuation phase fluoxetine
  Acute phase cognitive therapy : For the first 12 weeks, all participants received between 16 and 20 cognitive therapy sessions.
  Continuation phase fluoxetine : The dosage of fluoxetine was increased to 40 mg over 8 months.
Period: Overall Study
Arm/Group | Continuation Phase Fluoxetine | Continuation Phase Cognitive Therapy | Continuation Phase Pill Placebo
Started | 86 | 86 | 69
Completed | 62 | 70 | 49
Not Completed | 24 | 16 | 20

BASELINE CHARACTERISTICS:
Population: 523 adults with recurrent major depressive disorder began acute phase cognitive therapy; only the 241 eligible higher-risk responders were randomized to the 3 arms above.
Groups:
- Total: Total of all reporting groups
Arm/Group | Continuation Phase Fluoxetine | Continuation Phase Cognitive Therapy | Continuation Phase Pill Placebo | Total
Number analyzed (Participants) | 86 | 86 | 69 | 241
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 86 | 86 | 69 | 241
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.6 (11.8) | 43.1 (11.5) | 43.6 (12.3) | 42.7 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 63 | 42 | 162
  Male | 29 | 23 | 27 | 79
Region of Enrollment [Number; unit: participants]
  United States | 86 | 86 | 69 | 241

OUTCOME MEASURES:

1. Primary Outcome: Depressive Relapse or MDD
Description: Longitudinal Interval Follow-up Evaluation - Psychiatric Status Rating (LIFE-PSR) of 5 or more (on a scale from 1 to 6 measuring major depressive disorder) for 2 consecutive weeks according to evaluator blinded to randomized assignment
  LIFE-PSR Scale:
  1. = No residual symptoms, no current evidence of the disorder.
  2. = Mild symptoms
  3. = Considerably less psychopathology than full criteria with no more than moderate impairment
  4. = Does not meet full criteria but has major symptoms of impairment
  5. = Meets criteria without extreme impairment in functioning
  6. = Meets criteria with extreme impairment in functioning
  The relapse rate was estimated using Kaplan-Meier estimates (Kaplan, Meier J Am Stat, 1958, pp.457-481)
Time Frame: Measured at month 8
Population: Intention to treat analysis
Measure: Number; unit: % patients who relapsed
Arm/Group | Continuation Phase Fluoxetine | Continuation Phase Cognitive Therapy | Continuation Phase Pill Placebo
Number analyzed (Participants) | 86 | 86 | 69
% patients who relapsed | 18 | 18.3 | 32.7
Statistical Analysis 1: Comparison: Continuation Phase Fluoxetine vs Continuation Phase Cognitive Therapy; The sample size was based on a predicted 30% difference in relapse/recurrence rates between C-CT and fluoxetine (ie,30% vs 60%) across both the experimental phase and the first 12 months of follow-up. With these assumptions, 180 randomized patients (60 per cell) were required to detect a statistically significant difference using a log-rank test with 1-sided α = 0.05 and 80% power; Test type: Superiority or Other; p = .42, Log Rank; log-rank chi-square = 0.038, df = 1, p <=.42; Hazard Ratio (HR) = 1.079, 95% CI 2-sided [0.50 to 2.34], Standard Error of Mean .39 — Hazard ratio for relapse in C-CT group compared to that in the fluoxetine group
Statistical Analysis 2: Comparison: Continuation Phase Fluoxetine vs Continuation Phase Pill Placebo; Test type: Superiority or Other; p = .02, Log Rank; log-rank chi-square = 3.92, df = 1; Hazard Ratio (HR) = .481, 95% CI 2-sided [.23 to 1.01], Standard Error of Mean .38 — Hazard Ratio for relapse in fluoxetine group compared to that in the pill placebo group
Statistical Analysis 3: Comparison: Continuation Phase Cognitive Therapy vs Continuation Phase Pill Placebo; Test type: Superiority or Other; p = .03, Log Rank; log-rank chi-square = 3.391, df = 1; Hazard Ratio (HR) = 0.519, 95% CI 2-sided [0.26 to 1.06], Standard Error of Mean .36 — Hazard ratio for relapse in C-CT group compared to that in the placebo group
Statistical Analysis 4: Comparison: Continuation Phase Fluoxetine vs Continuation Phase Cognitive Therapy vs Continuation Phase Pill Placebo; Test type: Superiority or Other; p = .01, Log Rank; log-rank chi-square = 5.06, df = 1; Hazard Ratio (HR) = 0.501, 95% CI 2-sided [0.27 to 0.93], Standard Error of Mean .31 — Hazard ratio for relapse in active treatment group (fluoxetine or C-CT) compared to that in the placebo group

2. Primary Outcome: Depressive Relapse/Recurrence or MDD
Description: Longitudinal Interval Follow-up Evaluation - Psychiatric Status Rating (LIFE-PSR) of 5 or more (on a scale from 1 to 6 measuring MDD) for 2 consecutive weeks according to evaluator blinded to randomized assignment
  LIFE-PSR Scale:
  1. = No residual symptoms, no current evidence of the disorder.
  2. = Mild symptoms
  3. = Considerably less psychopathology than full criteria with no more than moderate impairment
  4. = Does not meet full criteria but has major symptoms of impairment
  5. = Meets criteria without extreme impairment in functioning
  6. = Meets criteria with extreme impairment in functioning
  Relapse/recurrence rate was estimated using Kaplan-Meier estimates (Kaplan, Meier J Am Stat, 1958, pp.457-481)
Time Frame: Measured at month 20
Population: Intention to treat analysis
Measure: Number; unit: % patients who relapsed/recurred
Arm/Group | Continuation Phase Fluoxetine | Continuation Phase Cognitive Therapy | Continuation Phase Pill Placebo
Number analyzed (Participants) | 86 | 86 | 69
% patients who relapsed/recurred | 35.1 | 35.0 | 42.7
Statistical Analysis 1: Comparison: Continuation Phase Fluoxetine vs Continuation Phase Cognitive Therapy; Test type: Superiority or Other; p = .48, Log Rank; log-rank chi-square = 0.002, df = 1; Hazard Ratio (HR) = 0.988, 95% CI 2-sided [0.55 to 1.76], Standard Error of Mean .30 — Hazard ratio for relapse/recurrence in the C-CT group compared to that in the fluoxetine group
Statistical Analysis 2: Comparison: Continuation Phase Fluoxetine vs Continuation Phase Pill Placebo; Test type: Superiority or Other; p = .14, Log Rank; Chi-square = 1.19, df = 1; Hazard Ratio (HR) = .717, 95% CI 2-sided [.39 to 1.31], Standard Error of Mean .31 — Hazard ratio of relapse/recurrence in the Fluoxetine arm over the 20 months of follow-up since randomization compared to the pill placebo arm
Statistical Analysis 3: Comparison: Continuation Phase Cognitive Therapy vs Continuation Phase Pill Placebo; Test type: Superiority or Other; p = .13, Log Rank; chi-square = 1.262, df = 1; Hazard Ratio (HR) = .715, 95% CI 2-sided [.40 to 1.29], Standard Error of Mean .30 — Hazard ratio of relapse/recurrence in the C-CT arm over the 20 months of follow-up since randomization compared to the pill placebo arm
Statistical Analysis 4: Comparison: Continuation Phase Fluoxetine vs Continuation Phase Cognitive Therapy vs Continuation Phase Pill Placebo; Test type: Superiority or Other; p = .10, Log Rank; Chi-square = 1.595, df = 1; Hazard Ratio (HR) = .717, 95% CI 2-sided [.43 to 1.20], Standard Error of Mean .26 — Hazard of relapse/recurrence in the active treatment (FLX or C-CT) arm compared to PBO (placebo)arm

3. Primary Outcome: Depressive Relapse/Recurrence or MDD
Description: as for outcome 2
Time Frame: Measured at month 32
Population: Intention to treat analysis
Measure: Number; unit: % patients who relapsed/recurred
Arm/Group | Continuation Phase Fluoxetine | Continuation Phase Cognitive Therapy | Continuation Phase Pill Placebo
Number analyzed (Participants) | 86 | 86 | 69
% patients who relapsed/recurred | 41.1 | 45.2 | 56.3
Statistical Analysis 1: Comparison: Continuation Phase Fluoxetine vs Continuation Phase Cognitive Therapy; Test type: Superiority or Other; p = .40, Log Rank; chi-square = .07, df = 1; Hazard Ratio (HR) = 1.075, 95% CI 2-sided [.63 to 1.84], Standard Error of Mean .27 — Hazard of relapse/recurrence for C-CT arm compared to FLX arm was reported
Statistical Analysis 2: Comparison: Continuation Phase Fluoxetine vs Continuation Phase Pill Placebo; Test type: Superiority or Other; p = .61, Log Rank; chi-square = 2.407, df = 1; Hazard Ratio (HR) = .649, 95% CI 2-sided [.37 to 1.13], Standard Error of Mean .28 — Hazard of relapse/recurrence in the FLX arm compared tp C-CT arm was reported
Statistical Analysis 3: Comparison: Continuation Phase Cognitive Therapy vs Continuation Phase Pill Placebo; Test type: Superiority or Other; p = .09, Log Rank; chi-square = 1.731, df = 1; Hazard Ratio (HR) = .701, 95% CI 2-sided [.41 to 1.19], Standard Error of Mean .27 — Hazard of relapse/recurrence in the C-CT arm compared to PBO arm is reported
Statistical Analysis 4: Comparison: Continuation Phase Fluoxetine vs Continuation Phase Cognitive Therapy vs Continuation Phase Pill Placebo; Test type: Superiority or Other; p = .05, Log Rank; chi-square = 2.705, df = 1; Hazard Ratio, log = .676, 95% CI 2-sided [.42 to 1.08], Standard Error of Mean .24 — Hazard of relapse/recurrence in the active treatment (FLX or C-CT) arm compared to PBO arm was reported

ADVERSE EVENTS:
Time Frame: 32 months
Arm/Group | Continuation Phase Fluoxetine | Continuation Phase Cognitive Therapy | Continuation Phase Pill Placebo
Serious Adverse Events (participants affected / at risk) | 0/86 | 0/86 | 0/69
Other Adverse Events (participants affected / at risk) | 0/86 | 0/86 | 0/69

LIMITATIONS AND CAVEATS:
To our knowledge in 2014 this is of the largest, cognitive therapy responders who presented with recurrent MDD and were followed longitudinally

Proficient therapists;competency measured.

Generalizability is limited by design characteristics.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No